CLINICAL TRIAL: NCT01878552
Title: Energy Load During Mechanical Ventilation in Patients With Acute Respiratory Distress Syndrome (ARDS)
Brief Title: Energy Load in Patients With Acute Respiratory Distress Syndrome (ARDS)
Status: Completed | Type: Observational
Sponsor: Policlinico Hospital (Other)
Responsible Party: Principal Investigator, Davide Chiumello, MD, Policlinico Hospital
Other Study IDs: Policlinico-07
Record Dates: First submitted 2013-06-07; First posted 2013-06-17 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Acute Respiratory Distress Syndrome (ARDS)
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ARDS: Mechanically ventilated patients with Acute Respiratory Distress Syndrome

SUMMARY:
The investigator would assess if there is an incremental energy load during mechanical ventilation in Acute Respiratory Distress Syndrome (ARDS) patients.

DETAILED DESCRIPTION:
The investigator would study the inspiratory and expiratory pressure volume curve in ARDS patients and investigate if there is a correlation between the energy loss (hysteresis curve) and the severity of disease.

ELIGIBILITY:
Inclusion Criteria:

* ARDS patients

Exclusion Criteria:

* pediatric population
* Chronic Obstructive Pulmonary Disease (COPD)
* patients with hemodynamic instability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ARDS patients
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2013-04; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Mortality | Two weeks (average ICU stay)
  Association between energy load provided to the lung during mechanical ventilation and mortality during ICU stay

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinico hospital, Mialn, Italy, Italy